CLINICAL TRIAL: NCT00551317
Title: A Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Single Oral Doses of Darapladib (SB480848) in Healthy Japanese Male Subjects
Brief Title: A Study Investigating the Concentrations of Darapladib in Blood and the Safety of This Compound in Healthy Japanese Men
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: LPL110077
Record Dates: First submitted 2007-10-29; First posted 2007-10-30 (Estimated); Last update posted 2016-12-05 (Estimated); Status verified 2016-12

CONDITIONS: Atherosclerosis
Keywords: SB480848,; Japanese healthy volunteers; darapladib,
MeSH Terms: conditions — Atherosclerosis | interventions — darapladib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Darapladib (SB480848)

SUMMARY:
This study is being conducted to provide initial safety, tolerability, PK and PD data that will allow further studies with darapladib in Japanese patients

ELIGIBILITY:
Inclusion criteria:

* Japanese males, 20-64 years of age, inclusive
* Body weight >50Kg
* Body Mass Index (BMI): 18-28
* Subjects must have lived outside of Japan no more than 10 years
* Non-smoker or smokes fewer than 10 cigarettes/day

Exclusion criteria:

* History of asthma, anaphylaxis or anaphylactoid reactions, severe allergic responses
* History of sensitivity to heparin or heparin-induced thrombocytopenia
* History of alcohol/drug abuse or dependence within 12 months of the study
* Positive syphilis, HIV antibody, Hepatitis B, Hepatitis C
* History of cholecystectomy or biliary tract disease or history of liver disease
* Participation in a clinical study within 30 days prior to first dose
* Subject has been exposed to more than 4 chemical entities within 12 months
* Positive urine drug and alcohol at screening
* Subject has any medical history or clinically relevant abnormality that would make the subject ineligible for inclusion due to safety reasons.

Ages: 20 Years to 64 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2007-07; Primary Completion 2007-09 (Actual); Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
- Safety/tolerability of single oral doses of darapladib | 4, 24 and 96h post-dose
- Primary Pharmacokinetic parameters of single oral doses of darapladib | pre-dose, 0,5, 1, 2, 3, 4, 6, 9 12, 16, 24, 48, 72h post-dose

SECONDARY OUTCOMES:
-Secondary PK parameters -PK parameters of SB553253 -inhibition of Lp-PLA2 activity -description of plasma concentration-Lp-PLA2 activity inhibition relationship after single oral doses of darapladib. all measured same timepoints as primary PK | Throughout the study

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Honolulu, Hawaii, United States

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Dataset Specification: LPL110077 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: LPL110077 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: LPL110077 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: LPL110077 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: LPL110077 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: LPL110077 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: LPL110077 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register